CLINICAL TRIAL: NCT06282302
Title: Effect of Isometric and Aerobic Physical Exercise on Blood Pressure Levels in Hypertensive Elderly People: Randomized Clinical Trial
Brief Title: Effect of Isometric and Aerobic Physical Exercise on Blood Pressure Levels in Hypertensive Elderly People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6030/22
Record Dates: First submitted 2024-01-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Hypertension,Essential; Hypertension
Keywords: hypertension; isometric exercise; aerobic exercise
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Control Groups; Exercise

STUDY DESIGN:
Intervention Model Description: The RCT will involve thirty-six elderly volunteers (≥ 60 years of age) with systemic arterial hypertension, aiming to compare two types of physical exercise sessions, isometric wall squats and an aerobic exercise session on an exercise bike, on the 24-hour blood pressure levels.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group control (Experimental): The control session will consist of keeping the volunteer sitting in a calm, air-conditioned environment for 40 minutes.
  Interventions: Other: Group control
- Isometric Exercise (Experimental): The intervention with isometric exercise for the lower limbs, the volunteers will start in a vertical position, with shoulders and hips in contact with the wall, feet parallel and shoulder-width apart and hands at the sides of the body. Then (second phase), the volunteers, maintaining contact with the wall, squatted and advanced their feet in the desired position until the knee joint angle reached the previously determined value. The third phase referred directly to the isometric effort of the isometric exercise session. For the isometric wall squat exercise session, volunteers will be asked to perform 4 repetitions of 2 minutes, with a 2-minute rest interval in a seated position for adequate rest between each repetition.
  Interventions: Other: Isometric Exercise
- Aerobic Exercise (Experimental): Volunteers will perform 50 minutes of horizontal exercise cycling (brand: pro-user), continuously and at moderate intensity (50% to 60% of HR reserve).
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Group control — Group control The control session will consist of keeping the volunteer sitting in a calm, air-conditioned environment for 40 minutes.
  Arms: Group control
Other: Isometric Exercise — The intervention with isometric exercise for the lower limbs, the volunteers will start in a vertical position, with shoulders and hips in contact with the wall, feet parallel and shoulder-width apart and hands at the sides of the body. Then (second phase), the volunteers, maintaining contact with the wall, squatted and advanced their feet in the desired position until the knee joint angle reached the previously determined value. The third phase referred directly to the isometric effort of the isometric exercise session. For the isometric wall squat exercise session, volunteers will be asked to perform 4 repetitions of 2 minutes, with a 2-minute rest interval in a seated position for adequate rest between each repetition.
  Arms: Isometric Exercise
Other: Aerobic Exercise — Volunteers will perform 50 minutes of horizontal exercise cycling (brand: pro-user), continuously and at moderate intensity (50% to 60% of HR reserve).
  Arms: Aerobic Exercise

SUMMARY:
Introduction: Adequate blood pressure control is necessary to reduce the risk of mortality from cardiovascular events. The effects of aerobic exercise on systemic arterial hypertension are already well known, however, to date, there is little evidence regarding the effect of an isometric exercise session for the lower limbs on blood pressure levels, especially when performed in elderly hypertensive individuals. Objective: To verify the effect of an isometric or aerobic exercise protocol for the lower limbs on 24-hour ambulatory blood pressure in elderly hypertensive individuals.

DETAILED DESCRIPTION:
Introduction: Adequate blood pressure control is necessary to reduce the risk of mortality from cardiovascular events. The effects of aerobic exercise on systemic arterial hypertension are already well known, however, to date, there is little evidence regarding the effect of an isometric exercise session for the lower limbs on blood pressure levels, especially when performed in elderly hypertensive individuals. Objective: To verify the effect of an isometric or aerobic exercise protocol for the lower limbs on 24-hour ambulatory blood pressure in elderly hypertensive individuals.

Methods: Thirty-six controlled hypertensive volunteers, aged ≥ 60 years, of both sexes, will be randomly selected based on their medical records. Volunteers will be randomized to perform an isometric wall squat exercise session (n=12 - 4 repetitions of 2 minutes of execution and 2 minutes of rest, performed at a specific angle of the volunteer's knee joint - Borg scale of 11 to 13 points - moderate intensity) or an aerobic exercise session on a stationary bike (n=12 - 40 minutes and at moderate intensity stipulated between the range of 50% to 60% of HR reserve and Borg scale of 11 to 13 points - moderate intensity) or a control session without exercise, 40 minutes per session (n=12). 24-hour Ambulatory Blood Pressure Monitoring will be performed pre- and post-session. Statistical analyzes will be performed using the ANOVA test (one way), power of 80% and alpha 95%, SPSS-26.0.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive elderly;
* Both genders;
* Aged ≥ 60 years;
* Hypertensive patients on continuous use of antihypertensive medication;
* Hypertensive who did not practice physical exercise regularly (≥ 2 sessions per week).

Exclusion Criteria:

* Those who presented one of the following issues will be excluded:
* Diabetes mellitus;
* Chronic renal failure;
* Body mass index (BMI) ≥ 35 kg/m2;
* Coronary artery disease;
* Heart failure;
* Any injury to the lower limbs;
* Smokers.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-03-18 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
24-hour Ambulatory Blood Pressure Monitoring | Until completion of the study, on average 4 months.
  Check 24-hour blood pressure levels (24-hour Ambulatory Blood Pressure Monitoring) obtained after an isometric squat session in elderly individuals with SAH and compare BP levels after an exercise session on a stationary bike and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: LIDIANE P STOCHERO, Principal Investigator — University Foundation of Cardiology
Locations (1):
- Institute of Cardiology, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Summary Study protocol Statistical Analysis Plan (SAP) Free and Informed Consent Form (TCLE) Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months
Access Criteria: University Foundation of Cardiology

REFERENCES:
- [Background] Oliveira PC, Silva MR, Lehnen AM, Waclawovsky G. Isometric handgrip training, but not a single session, reduces blood pressure in individuals with hypertension: a systematic review and meta-analysis. J Hum Hypertens. 2023 Sep;37(9):844-853. doi: 10.1038/s41371-022-00778-7. Epub 2022 Nov 15. PMID 36379974
- [Background] Saco-Ledo G, Valenzuela PL, Ramirez-Jimenez M, Morales JS, Castillo-Garcia A, Blumenthal JA, Ruilope LM, Lucia A. Acute Aerobic Exercise Induces Short-Term Reductions in Ambulatory Blood Pressure in Patients With Hypertension: A Systematic Review and Meta-Analysis. Hypertension. 2021 Dec;78(6):1844-1858. doi: 10.1161/HYPERTENSIONAHA.121.18099. Epub 2021 Nov 1. PMID 34719262
- [Background] Pescatello LS, Franklin BA, Fagard R, Farquhar WB, Kelley GA, Ray CA; American College of Sports Medicine. American College of Sports Medicine position stand. Exercise and hypertension. Med Sci Sports Exerc. 2004 Mar;36(3):533-53. doi: 10.1249/01.mss.0000115224.88514.3a. PMID 15076798
- [Background] Waclawovsky G, Pedralli ML, Eibel B, Schaun MI, Lehnen AM. Effects of Different Types of Exercise Training on Endothelial Function in Prehypertensive and Hypertensive Individuals: A Systematic Review. Arq Bras Cardiol. 2021 May;116(5):938-947. doi: 10.36660/abc.20190807. English, Portuguese. PMID 34008818
- [Background] Pescatello LS, Bairos L, Vanheest JL, Maresh CM, Rodriguez NR, Moyna NM, DiPasquale C, Collins V, Meckes CL, Krueger L, Thompson PD. Postexercise hypotension differs between white and black women. Am Heart J. 2003 Feb;145(2):364-70. doi: 10.1067/mhj.2003.107. PMID 12595857
- [Background] Pescatello LS, Kulikowich JM. The aftereffects of dynamic exercise on ambulatory blood pressure. Med Sci Sports Exerc. 2001 Nov;33(11):1855-61. doi: 10.1097/00005768-200111000-00009. PMID 11689735
- [Background] Baross AW, Wiles JD, Swaine IL. Double-leg isometric exercise training in older men. Open Access J Sports Med. 2013 Jan 30;4:33-40. doi: 10.2147/OAJSM.S39375. eCollection 2013. PMID 24379707
- [Background] Ash GI, Taylor BA, Thompson PD, MacDonald HV, Lamberti L, Chen MH, Farinatti P, Kraemer WJ, Panza GA, Zaleski AL, Deshpande V, Ballard KD, Mujtaba M, White CM, Pescatello LS. The antihypertensive effects of aerobic versus isometric handgrip resistance exercise. J Hypertens. 2017 Feb;35(2):291-299. doi: 10.1097/HJH.0000000000001176. PMID 27861249